CLINICAL TRIAL: NCT06265168
Title: Comprehensive Observations and Multidisciplinary Approaches in the Management of Unconscious Patients - a Prospective High Fidelity Simulator Study
Brief Title: Comprehensive Observations and Multidisciplinary Approaches in the Management of Unconscious Patients
Acronym: COMA
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: req-2023-01512; am23Sutter3
Record Dates: First submitted 2024-02-05; First posted 2024-02-20 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Coma
Keywords: high-fidelity simulation; observational study
MeSH Terms: conditions — Coma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians: Volunteering intensivists, emergency physicians, internists, and neurologists.
  Interventions: Other: Simulation

INTERVENTIONS:
Other: Simulation — Physicians will participate in a simulated scenario of an adult comatose patient. The intervention will be presented as a learning situation where the physician interacts with a high-fidelity mannequin. The mannequin simulating the patient will manifest a Glasgow Coma Score of 3 (improving over time to a GCS of 4) and a range of physiological and pathological symptoms. Physicians will have access to emergency equipment, including intubation equipment, a defibrillator, and medications. A trained nurse will be present to assist with the simulation. After 20 minutes the patient will regain consciousness in order to avoid a frustrating experience for the physicians. After simulation termination, a senior physician will join the resident and ask him to report the current scenario and will stop the simulation. The entire scenario will be video-recorded.

SUMMARY:
This prospective observational high-fidelity simulation study aims to observe and better understand how physicians from different disciplines differentiate in the management of a comatose patient and how their diagnostic and treatment approaches adhere to current recommendations in a highly standardized simulated scenario. The results gained by this study will give more insight into the current quality of diagnostic procedures and treatment and help refine recommendations in this context. The investigators hypothesize that physicians do not strictly adhere (regarding diagnostic approach and treatment) to current guidelines/recommendations when confronted with a comatose patient.

DETAILED DESCRIPTION:
Each participant will attend one study visit. For all participants, the investigators will offer an emergency high-fidelity simulator training workshop. The study will be presented as a learning situation, in which the participating physicians can train and improve their skills in medical emergencies. All participating physicians will be asked to complete two questionnaires (one before and one after the simulation). The first includes questions about age, medical knowledge, medical specialization, prior experience with simulator-based training, clinical experience, hours worked prior to simulation and their stress level (quantified as 0 [not stressed] and 10 [severely stressed]).

All physicians will be informed regarding the features of the high-fidelity mannequin (see respective subjection below), the equipment of the artificial emergency room, and the role of a resident in the emergency department. The second questionnaire will include questions aimed at understanding the clinical experience, knowledge, and conceptual understanding regarding diagnostics and management of coma. The simulation will be terminated after 20 minutes. All physicians will be exposed to the scenario once (the clinical case is detailed in the respective subjection below).

No information about the workshop's goal or the scenarios' content will be given to the physicians before the simulation. After the simulation, the physicians will be asked to perform a short self-assessment using an "emotion wheel simulation reflexivity" questionnaire.

The mannequin can talk, blink, open or close eyes and mouth, produce foamy sputum, enuresis, and move the pupils and extremities symmetrically or asymmetrically. The pupils can be reactive or unreactive to light. Pulses can be palpated, thoracic excursion and pulmonary sounds during breathing can be detected. The vital signs (including breathing frequency, heart rate, oxygenation, and blood pressure) and the electrocardiogram of the mannequin are displayed on a standard monitoring device at bedside. The simulator room will be equipped with a manual external defibrillator, standard emergency medications (including Vasopressors, Steroids, Antimicrobials, crystalloid fluid, Glucose-infusions etc), intubation equipment, suctioning tubes, bandages, a pocket flashlight (to check pupils) and a stethoscope. A printed version of the medical chart will contain a written report of the emergency medical service and laboratory results (including blood gas analysis and hemogram revealing normal values, normoglycemia, normal C-reactive protein serum concentration, normal thyroid-stimulating hormone levels, negative routine toxicologic screening results, elevated liver enzyme serum levels, normal measures of cerebrospinal fluid analysis, and an increased osmotic gap which will only be presented upon request of the physician). During the scenario, the programmed measures of vital signs of the mannequin (including breathing frequency, heart rate, oxygenation, and blood pressure) and their changes over time will be displayed on a standard bedside monitoring device and present normal values. An unremarkable cerebral computed tomogram will be displayed. An intravenous access will be pre-installed for the application of medications or fluids. During the simulation, a trained critical care study nurse (confederate) will be present to support the physician regarding the ascertainment of diagnostic results, attaching and initiating monitoring devices, and preparation. The study nurse is trained not to instruct physicians about the diagnostic workup or to reveal treatment algorithms and will administer drugs only at the physician's demand. The use of electronic devices to access institutional or international guidelines and literature is permitted. The entire scenario will be monitored by a mobile camera and microphone allowing simultaneous video and audio recording of the team performance and monitor findings. The recording will also be used for debriefing purposes and (if consent is given by the physician) for anonymized analyzes regarding the study aims. Debriefing sessions will be conducted individually after each training.

ELIGIBILITY:
Inclusion Criteria:

* The participant is a physician (one of the following specialties: Neurology, Intensive Care, Internal Medicine, Emergency Medicine)
* The participant practices medicine at the University Hospital Basel
* The participant has signed informed consent and agrees to be recorded (audio and video) during the study.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Physicians from different medical specialties (including neurologists, intensivists, internists, and emergency medical doctors) with different duration of clinical experience working at the University Hospital Basel.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To reveal diagnostic and treatment approaches of physicians from different disciplines when confronted with a comatose patient. | 1 time assessment before, during and directly after the intervention (approx. 30 minutes in total)

SECONDARY OUTCOMES:
Physicians' grade of adherence to current recommendations regarding diagnostic procedures and treatment of a comatose patient | 1 time assessment during and directly after the intervention (approx. 30 minutes in total)
Participants' self-evaluation of their performance in hindsight | 1 time assessment directly after the intervention (approx. 10 minutes in total)

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liliane N, Tisljar K, Berger S, De Marchis GM, Dittrich TD, Bassetti S, Bingisser R, Hunziker S, Marsch S, Sutter R. Comprehensive observations and multidisciplinary approaches (COMA) in the management of unconscious patients: a prospective high fidelity simulation study. J Neurol. 2025 Jul 25;272(8):537. doi: 10.1007/s00415-025-13228-4. PMID 40711621